CLINICAL TRIAL: NCT05942794
Title: Use of a Tissue Autofluorescence Detection System for Identification of Oral Mucosal Lesions
Brief Title: Identification of Oral Lesions Through an Autofluorescence System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Luca Ramaglia, Clinical Professor, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 177/2023
Record Dates: First submitted 2023-06-29; First posted 2023-07-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Oral Leukoplakia; Autofluorescence; Secondary Prevention; Keratosis; Oral Lichen Planus; Oral Cancer; Oral Disease
Keywords: Oral Leukoplakia; Lichen Planus; Squamous cell carcinoma; Keratosis
MeSH Terms: conditions — Leukoplakia, Oral; Keratosis; Lichen Planus, Oral; Mouth Neoplasms; Mouth Diseases; Lichen Planus; Carcinoma, Squamous Cell

STUDY DESIGN:
Intervention Model Description: The screening will start after a first oral examination, in order to rule out noticeable mucosal lesions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening examination (Experimental): All patients will undergo a screening examination (with or without GOCCLES ® glasses) by all three operators.
  Interventions: Device: Screening examination

INTERVENTIONS:
Device: Screening examination — After an initial clinical visit, all three operators will wear the tissue autofluorescence detection device (GOCCLES®), reporting both observations on their "operator-module".

SUMMARY:
The aim of the study will be to evaluate the efficacy of a tissue autofluorescence detection system as an aid to clinical screening in identifying lesions of the oral mucosa. The screening process will be performed by 3 clinicians with a different level of experience. Sensitivity and specificity tests will be conducted.

DETAILED DESCRIPTION:
Tissue autofluorescence analysis will be performed using GOOCLES® glasses, a device capable of detecting variations in fluorescence when the examined area is illuminated with a common photopolymerising lamp. Three clinical professionals will be identified:

* Dental hygienist (1);
* General dentist (2);
* Dentist expert in Medicine and Oral Pathology (3).

All patients will be included in the study after receiving an initial dental visit, in order to rule out patients with noticeable oral lesions.

Dental hygienist (1) will collect the patient's data by filling the "anamnestic record". Furthermore, (1) will perform the first clinical examination (with and without GOOCLES®), reporting his observations on his own "operator module".

The same screening (with and without GOOCLES®) will be conducted blindly by the general dentist (2) who, if he deems it necessary, will refer the patient to the oral pathologist (3), who will confirm or not (with and without GOOCLES®) the presence of an oral region such as to be further investigated (follow up or biopsy) and will report the observations on its own "operator module".

Inter-operator and intra-operator comparisons will be performed and the data thus obtained will be processed for statistical processing.

ELIGIBILITY:
Inclusion Criteria:

* Male and female;
* Age ≥ 18 years;
* Non-smokers and smokers

Exclusion Criteria:

* Cancer patients;
* Patients presenting a histological diagnosis of oral mucosal dysplasia/carcinoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical change of oral mucosa | baseline and after 21 days
  Presence of a white, red, or mixed mucosal area with an exophytic or vegetative appearance or with loss of substance
Fluorescence change of oral mucosa | baseline and after 21 day
  Presence of a mucosal area with reduced or increased fluorescence

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No